CLINICAL TRIAL: NCT05560425
Title: Pilot Study on Mindfulness Meditation and Behavioral Flexibility Among Emerging Adults
Brief Title: Pilot Study on Training Emerging Adults Skills in Navigating College
Acronym: SINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21-1486
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Abuse; Cognitive Deficit in Attention
Keywords: Attentional Bias; Alcohol Misuse; Emerging Adults; Mindfulness Meditation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: parallel assignment randomized controlled trial feasibility study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigating College (NC) Training (Active Comparator): Control Group
  Interventions: Behavioral: Navigating College (NC) Training
- Koru Mindfulness (KM) Training (Experimental): Study Group
  Interventions: Behavioral: Koru Mindfulness (KM) Training

INTERVENTIONS:
Behavioral: Koru Mindfulness (KM) Training — The Koru Basic curriculum consists of four weekly interactive 75-minute classes delivered online through Zoom. Each class consists of an overview of 2-3 skills, group practice of the skills, and group reflection. Topics discussed during each training visit include: belly breathing, dynamic breathing, body scan (week 1); walking meditation, gatha (week 2); guided imagery, labeling thoughts (week 3); eating meditation, and labeling feelings (week 4). Participants are instructed to practice a skill for 10 minutes/day and log any reflection on that practice using the Koru phone application.
  Other Names: Koru Basic
  Arms: Koru Mindfulness (KM) Training
Behavioral: Navigating College (NC) Training — With topics discussed from the Freshman Survival Guide book, this training provides a closely matched active control group for KM Training. The training consists of four weekly 75-minute classes delivered online through Zoom. Each class consists of lecture and group discussions on topics related to navigating college. Topics discussed during each training visit include: habits, roommate issues, homesickness, the internet (week 1); strategies when sinking, study skills, getting involved, habit formation (week 2); HALT, gateway habit (week 3); and academic success tips, taking notes, and procrastination (week 4). Participants are instructed to journal about learned information and skills for 10 minutes/day.
  Arms: Navigating College (NC) Training

SUMMARY:
Lifetime risk for developing an alcohol use disorder increases with earlier onset of alcohol consumption. This risk may reflect a tendency for escalated alcohol intake among youth due to immature executive control, leading to more frequent binge drinking, which is associated with more alcohol-related problems. Binge drinking is associated with deficits in behavioral flexibility, which may suggest impaired control networks that contribute to automatic behavior. Individuals with an alcohol or substance use disorder (A/SUD) exhibit attentional bias toward drug- or alcohol-related stimuli that have attained salience through consistent use. Reward history increases attention towards non-drug stimuli, even among individuals with no lifetime A/SUD. Preliminary data (from Dr. Boettiger's lab) from a nationally representative US adult sample using data collected via Prolific found that a questionnaire measure of mindfulness moderates the relationship between alcohol misuse and attention to reward. Given evidence that heavy alcohol drinking impairs behavioral flexibility, which in turn promotes escalating intake, insight into the relationship between mindfulness and behavioral flexibility could inspire new strategies to prevent alcohol and substance use disorders in people at elevated risk.

DETAILED DESCRIPTION:
This is a feasibility pilot study of training freshman college students, with a history of alcohol binge drinking, mindfulness and meditation skills in 4 virtual visits. Before and after the virtual intervention, behavioral flexibility will be measured using a reward-driven attentional bias (Reward-AB) computerized task, and C-reactive protein (CRP) levels will be collected.

Upon arrival for the first visit, participants will be screened for any current alcohol intoxication or recent substance use, followed by a mental health assessment with the Mini-International Neuropsychiatric Interview (MINI). The participant will then have blood collected by finger prick, complete a Reward-AB task, and fill out some paper surveys. During visits 2 through 5, participants will complete virtual training on either mindfulness and meditation skills, or navigating college skills. Each visit will last approximately 90 minutes, starting with the completion of a few online surveys. Visit 6 is similar to visit 1, without the health interview. Participants will be contacted one month following the date of the 6th study visit to complete online surveys.

Visit 1:

* Written consent, MINI interview, urine drug screen and breathalyzer alcohol test, CRP assay, Reward-AB task.
* Randomization to either the Koru Mindfulness (KM) intervention or the Navigating College (NC) control group.

Visits 2-5:

* Surveys completed online through REDCap.
* 75 minutes of instructor-led discussion
* Breakout sessions for participants to share thoughts and experiences in response to instructor's prompt.

Visit 6:

Similar to visit 1, without repeating the MINI interview.

Follow-up:

One month after the conclusion of visit 6, participants will be contacted via email with a link to REDCap to complete several surveys.

Reward-Attentional Bias (Reward-AB) Task:

This computerized task will be used to measure attentional bias pre- and post-intervention. The task includes a training and testing portion, each of which are adapted from tasks that measure the influence of reward on visual attention.

Navigating College (NC) Control Group Training:

Topics discussed during each training visit include: habits, roommate issues, homesickness, the internet (week 1); strategies when sinking, study skills, getting involved, habit formation (week 2); Hungry, Angry, Lonely, and Tired (HALT), gateway habit (week 3); and academic success tips, taking notes, and procrastination (week 4).

Koru Mindfulness (KM) Intervention Training:

Topics discussed during each training visit include: belly breathing, dynamic breathing, body scan (week 1); walking meditation, gatha (week 2); guided imagery, labeling thoughts (week 3); eating meditation, and labeling feelings (week 4).

Daily Logging of Skills:

Participants in the NC intervention will be asked to journal by hand or via Qualtrics every day for >10 minutes, on anything related to the topics learned during that week's training visit. Participants in the KM intervention will be asked to practice every day for >10 minutes any mindfulness or meditation skill previously learned during training visits, in addition to logging practice of skills and reflection on the experience using the Koru application.

ELIGIBILITY:
Inclusion Criteria:

* High school educated; college enrolled first-year student
* Medically healthy
* Ages 18-19
* Native-English speaker (or fluent < 7 years old)
* Self-report of >4 lifetime binge drinking episodes (>4 drinks/2hours for females, >5 drinks/2 hours for males).

Exclusion Criteria:

* Psychiatric disease (such as depression or psychosis) using the MINI [25]
* Systemic disease such as cancer, cardiovascular or inflammatory disease which could influence cognitive functioning
* Motor or visual disturbance (e.g., colorblind)
* Current use of psychoactive drugs (aside from moderate caffeine or alcohol), including prescription medications, or individuals with a known history of any substance use disorders (not including alcohol; including nicotine) or desire to seek treatment for excess substance (not including alcohol) use.

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Boettiger, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Spear LP. Effects of adolescent alcohol consumption on the brain and behaviour. Nat Rev Neurosci. 2018 Apr;19(4):197-214. doi: 10.1038/nrn.2018.10. Epub 2018 Feb 15. PMID 29467469
- [Background] Mehrabian A, Russell JA. A questionnaire measure of habitual alcohol use. Psychol Rep. 1978 Dec;43(3 Pt 1):803-6. doi: 10.2466/pr0.1978.43.3.803. No abstract available. PMID 740823
- [Background] Gass JT, Glen WB Jr, McGonigal JT, Trantham-Davidson H, Lopez MF, Randall PK, Yaxley R, Floresco SB, Chandler LJ. Adolescent alcohol exposure reduces behavioral flexibility, promotes disinhibition, and increases resistance to extinction of ethanol self-administration in adulthood. Neuropsychopharmacology. 2014 Oct;39(11):2570-83. doi: 10.1038/npp.2014.109. Epub 2014 May 13. PMID 24820536
- [Background] Sey NYA, Gomez-A A, Madayag AC, Boettiger CA, Robinson DL. Adolescent intermittent ethanol impairs behavioral flexibility in a rat foraging task in adulthood. Behav Brain Res. 2019 Nov 5;373:112085. doi: 10.1016/j.bbr.2019.112085. Epub 2019 Jul 15. PMID 31319133
- [Background] Chanon VW, Sours CR, Boettiger CA. Attentional bias toward cigarette cues in active smokers. Psychopharmacology (Berl). 2010 Oct;212(3):309-20. doi: 10.1007/s00213-010-1953-1. Epub 2010 Jul 29. PMID 20668841
- [Background] Field M, Marhe R, Franken IH. The clinical relevance of attentional bias in substance use disorders. CNS Spectr. 2014 Jun;19(3):225-30. doi: 10.1017/S1092852913000321. Epub 2013 May 13. PMID 23663386
- [Background] Field M, Werthmann J, Franken I, Hofmann W, Hogarth L, Roefs A. The role of attentional bias in obesity and addiction. Health Psychol. 2016 Aug;35(8):767-80. doi: 10.1037/hea0000405. PMID 27505196
- [Background] Masiero M, Lucchiari C, Maisonneuve P, Pravettoni G, Veronesi G, Mazzocco K. The Attentional Bias in Current and Former Smokers. Front Behav Neurosci. 2019 Jul 10;13:154. doi: 10.3389/fnbeh.2019.00154. eCollection 2019. PMID 31354446
- [Background] Meyer KN, Sheridan MA, Hopfinger JB. Reward history impacts attentional orienting and inhibitory control on untrained tasks. Atten Percept Psychophys. 2020 Nov;82(8):3842-3862. doi: 10.3758/s13414-020-02130-y. PMID 32935290
- [Background] Greeson JM, Juberg MK, Maytan M, James K, Rogers H. A randomized controlled trial of Koru: a mindfulness program for college students and other emerging adults. J Am Coll Health. 2014;62(4):222-33. doi: 10.1080/07448481.2014.887571. PMID 24499130
- [Background] Anderson BA, Laurent PA, Yantis S. Value-driven attentional capture. Proc Natl Acad Sci U S A. 2011 Jun 21;108(25):10367-71. doi: 10.1073/pnas.1104047108. Epub 2011 Jun 6. PMID 21646524
- [Background] Anderson BA, Kim H, Britton MK, Kim AJ. Measuring attention to reward as an individual trait: the value-driven attention questionnaire (VDAQ). Psychol Res. 2020 Nov;84(8):2122-2137. doi: 10.1007/s00426-019-01212-3. Epub 2019 Jun 12. PMID 31190092
- [Background] Carmody J, Baer RA. Relationships between mindfulness practice and levels of mindfulness, medical and psychological symptoms and well-being in a mindfulness-based stress reduction program. J Behav Med. 2008 Feb;31(1):23-33. doi: 10.1007/s10865-007-9130-7. Epub 2007 Sep 25. PMID 17899351

RESULTS

PARTICIPANT FLOW:
Groups:
- Navigating College (NC) Training (Control Group): With topics discussed from the Freshman Survival Guide book, this training provides a closely matched active control group for KM Training. The training consists of four weekly 75-minute classes delivered online through Zoom. Each class consists of lecture and group discussions on topics related to navigating college. Topics discussed during each training visit include: habits, roommate issues, homesickness, the internet (week 1); strategies when sinking, study skills, getting involved, habit formation (week 2); Hungry, Angry, Lonely, Tired (HALT), gateway habit (week 3); and academic success tips, taking notes, and procrastination (week 4). Participants are instructed to journal about learned information and skills for 10 minutes/day.
- Koru Mindfulness (KM) Training (Study Group): The Koru Basic curriculum consists of four weekly interactive 75-minute classes delivered online through Zoom. Each class consists of an overview of 2-3 skills, group practice of the skills, and group reflection. Topics discussed during each training visit include: belly breathing, dynamic breathing, body scan (week 1); walking meditation, gatha (week 2); guided imagery, labeling thoughts (week 3); eating meditation, and labeling feelings (week 4). Participants are instructed to practice a skill for 10 minutes/day and log any reflection on that practice using the Koru phone application.
Period: Overall Study
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
Started | 7 | 9
Completed | 7 | 7
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: All 7 participants completed the NC Training, and 7 out of 9 participants completed the KM Training.
Groups:
- Navigating College (NC) Training (Control Group): With topics discussed from the Freshman Survival Guide book, this training provides a closely matched active control group for KM Training. The training consists of four weekly 75-minute classes delivered online through Zoom. Each class consists of lecture and group discussions on topics related to navigating college. Topics discussed during each training visit include: habits, roommate issues, homesickness, the internet (week 1); strategies when sinking, study skills, getting involved, habit formation (week 2); HALT, gateway habit (week 3); and academic success tips, taking notes, and procrastination (week 4). Participants are instructed to journal about learned information and skills for 10 minutes/day.
- Total: Total of all reporting groups
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group) | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.25 (0.38) | 18.00 (0) | 18.06 (0.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 4 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Participant Retention
Description: Participant retention will be measured by the percentage of enrolled participants remaining in the study after 6 visits.
Time Frame: 10 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
Number analyzed (Participants) | 7 | 9
percentage of participants | 85.71 | 88.89

2. Primary Outcome: Compliance With Independent Training of Skills
Description: To determine participant compliance with training skills learned during each of the 4 virtual visits, the average number of journal entries logged during the 4 weeks of training, for each group, is calculated as a total score (6 times/week x 4 weeks = 24). Scores range from 0 to 24, with higher scores indicating greater compliance with independent training.
Time Frame: 6 weeks
Population: Only 7 out of 9 participants in the KM Training group were analyzed because two participants dropped out of the study prior to completing the full duration of the training.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
Number analyzed (Participants) | 7 | 7
score on a scale | 10.43 (6.70) | 9.14 (6.18)
Statistical Analysis 1: Comparison: Navigating College (NC) Training (Control Group) vs Koru Mindfulness (KM) Training (Study Group); Null hypothesis: Compliance with independent training of skills is not equivalent between groups; Test type: Equivalence — The equivalence margin is a range of the compliance score for which the independent training of skills in each group is "close enough" to be considered equivalent; p < 0.05, t-test, 1 sided; degrees of freedom = 12; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-6.22 to 8.79], Standard Error of Mean 3.45

3. Secondary Outcome: Average CEQ Ratings - Credibility Subscale
Description: The Credibility subscale of the Credibility/Expectancy Questionnaire (CEQ) measures the the credibility of an intervention in clinical studies. The word "therapy" is replaced with "intervention" and modified to reflect the intent of the intervention (i.e., to improve skills in navigating college). Three items are each scored on a range from 0-9 and averaged together for a credibility rating, with high scores indicating greater perceived credibility of the intervention.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
Number analyzed (Participants) | 7 | 9
score on a scale | 15.29 (2.50) | 13.44 (2.70)

4. Secondary Outcome: Average CEQ Ratings - Expectancy Subscale
Description: The Expectancy subscale of the Credibility/Expectancy Questionnaire (CEQ) measures the the expectancy of an intervention in clinical studies. The word "therapy" is replaced with "intervention" and modified to reflect the intent of the intervention (i.e., to improve skills in navigating college). Three items are each scored on a range from 0-9 and averaged together for an expectancy rating, with high scores indicating greater perceived expectancy of positive outcomes of the intervention.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
Number analyzed (Participants) | 7 | 9
score on a scale | 13.29 (7.25) | 14.00 (5.34)

5. Secondary Outcome: Mean Change in Emotional Distress Scores
Description: The Depression, Anxiety and Stress Scale-21 (DASS-21) is composed of three self-report scales that measure depression, anxiety and stress. Items are rated on a Likert-type scale (0=Did not apply to me at all, to 3=Applied to me very much, or most of the time). Scores for the three subscales are calculated by summing the scores for the relevant items. The severity rating for Depression are Normal: 0-4, Mild: 5-6, Moderate: 7-10, Severe: 11-13, and Extremely Severe: 14-21; for Stress the ratings are Normal: 0-7, Mild: 8-9, Moderate: 10-12, Severe: 13-16, and Extremely Severe 17-21; and for Anxiety the ratings are Normal: 0-3, Mild: 4-5, Moderate: 6-7, Severe: 8-9, and Extremely Severe: 10-21. The total DASS-21 score is calculated by summing all three subscales, with a range from 0-63. For all scales, higher scores indicate greater emotional distress.
Time Frame: Baseline, Week 6
Population: Change scores could not be calculated for all participants for each subscale in the Navigating College (NC) Training (Control Group) due to missing data. Week 6 data were not collected for 2 participants in the Koru Mindfulness (KM) Training (Study Group).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
Number analyzed (Participants) | 7 | 7
score on a scale
  DASS-21 Total score: number analyzed (Participants) | 5 | 7
  DASS-21 Total score | 8.8 (7.1) | 4.6 (6.0)
  DASS-21 Depression score: number analyzed (Participants) | 6 | 7
  DASS-21 Depression score | 3.2 (2.9) | 2.6 (2.5)
  DASS-21 Anxiety score | 2.4 (0.6) | 0.6 (3.0)
  DASS-21 Stress score: number analyzed (Participants) | 6 | 7
  DASS-21 Stress score | 3.2 (2.1) | 1.4 (1.8)

6. Secondary Outcome: Participant Satisfaction
Description: Feedback will be collected the same day as each training visit, using a simple survey designed on Qualtrics.
Time Frame: 5 weeks
Population: Due to the time commitment burden on participants, data were not collected for this outcome.
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent at Visit 1 through the end of the study, a total of approximately 10 weeks.
Arm/Group | Navigating College (NC) Training (Control Group) | Koru Mindfulness (KM) Training (Study Group)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/25/NCT05560425/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT05560425/ICF_000.pdf